CLINICAL TRIAL: NCT06567847
Title: Is a Neurocognitively Enriched Exercise Effective in Reducing Re-Injury Risk and Improving Balance and Proprioception in Individuals With Lateral Ankle Instability?
Brief Title: Neurocognitive Exercises for Ankle Instability
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Collaborators: Bezmialem Vakif University (Other); Acıbadem Atunizade Hospital (Other)
Responsible Party: Principal Investigator, Aysenur Erekdag, Principal Investigator, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024_AE_Tez
Record Dates: First submitted 2024-08-20; First posted 2024-08-23 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Ankle Sprains
Keywords: Neuroplasticity; Reinjury; Chronic ankle instability; Physiotherapy
MeSH Terms: conditions — Ankle Injuries; Reinjuries

STUDY DESIGN:
Intervention Model Description: There will be an equal number of participants in the two groups randomized by the computer.
Who Masked: Outcomes Assessor
Masking Description: The assessor will not know which participant received which intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neurocognitive Enriched Exercise (Active Comparator): Individuals with a diagnosis of lateral ankle instability who underwent supervised neurocognitive enriched exercise under the guidance of a physiotherapist for 8 weeks, 2 days a week.
  Interventions: Other: Neurocognitive Enriched Exercise
- Multimodal Exercise (Active Comparator): Individuals with a diagnosis of lateral ankle instability who underwent supervised routine exercise under the guidance of a physiotherapist for 8 weeks, 2 days a week.
  Interventions: Other: Multimodal Exercise

INTERVENTIONS:
Other: Neurocognitive Enriched Exercise — An intervention planned, progressed, and conducted under the supervision of a physiotherapist, which enriches strengthening, balance, range of motion, stretching, and mobilization exercises with neurocognitive elements.
  Arms: Neurocognitive Enriched Exercise
Other: Multimodal Exercise — Supervised and progressively advanced interventions that include strengthening, balance, range of motion, stretching, and mobilization exercises.
  Arms: Multimodal Exercise

SUMMARY:
In the general population, 19.0-26.6 per 1000 cases of ankle instability have been reported, while in the athletic population, the rate is 11.3 per 1000. Ankle instability also predisposes individuals to recurrent instability, leading to persistent symptoms. After ankle injuries, temporary increases in afferent activity, along with long-term deficits in somatosensory information from ligaments, may cause central neuroplasticity that affects sensorimotor function. This central neuroplasticity can lead to permanent dysfunctions in the affected limb, thereby increasing the likelihood of developing and maintaining chronic ankle instability (CAI). In addition to the association between impaired balance and reduced proprioception with CAI, it has been reported that the central nervous system may fail to manage joint stress due to its inability to discern load on the ligaments.

Impaired neurocognition has been linked to decreased performance and higher rates of re-injury. Deficiencies in neuromuscular control, motor learning, or other neurocognitive components related to an individual's performance and safety may affect the ability to respond appropriately in a dynamic environment. Any deficiencies in these neurocognitive processes can hinder the successful completion of tasks.

The aim of this study is to comparatively examine the effects of neurocognitively enriched rehabilitation versus traditional rehabilitation on re-injury risk, balance, and proprioception in individuals with a history of ankle instability.

DETAILED DESCRIPTION:
Voluntary participants who have been diagnosed with lateral ankle instability will be included in the study. Signed voluntary consent will be obtained from participants. Participants will be divided into two groups. Study groups will be as follows: a) Neurocognitive Enriched Exercise, b) Multimodal Exercise.

ELIGIBILITY:
Inclusion Criteria:

* The documented unilateral ankle instability confirmed through clinical examinations (drawer test, talar tilt test) and MRI in cases requiring differential diagnosis.
* A history of an initial ankle sprain occurring at least 6 months ago.
* The presence of a recurrent sense of giving way that started at least 6 months ago and has been intermittently persistent.

Exclusion Criteria:

* Presence of a history of previous surgery in the lower extremity.
* Identification of organic and non-organic lesions such as cartilage injuries, periarticular tendon tears, and impingement syndromes.
* The existence of a fracture accompanying instability in the foot-ankle.
* Presence of congenital deformities in the foot-ankle.
* Diagnosis of talus osteochondral lesion.
* Diagnosis of ankle arthritis.
* Presence of medial ligament lesion.
* Existence of peripheral neuropathy.
* Presence of additional rheumatological diseases.
* Regular moderate-level exercise for at least 3 days a week in the last 6 months.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2027-11 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Cumberland Ankle Instability Tool (CAIT) | change from baseline at 6 months
  It is a 30-point, 9-item scale measuring the severity of functional ankle instability. Lower scores indicate functional ankle instability. The Minimal Clinically Important Difference for this valid and reliable scale is 3 points.
Surface Electromyography-maximum voluntary isometric contraction | change from baseline at 6 months
  Electrode placements will be performed in accordance with the European Recommendations from Surface EMG for Non-Invasive Assessment of Muscles (SENIAM).
Surface Electromyography-muscles' normal functional activities | change from baseline at 6 months
  Electrode placements will be performed in accordance with the European Recommendations from Surface EMG for Non-Invasive Assessment of Muscles (SENIAM).

SECONDARY OUTCOMES:
Ultrasonography | 3 times for 24 weeks
  The pennation angles of the peroneal, gastrocnemius, and tibialis anterior muscle groups will be evaluated and recorded using ultrasonographic imaging. The pennation angle will be defined as the angle between the muscle fascicle and the superficial aponeurosis.
Numeric Pain Rating Scale | 3 times for 24 weeks
  Pain during activity in the ankle will be assessed with a pain NPRS, a numbered scale of 11 points. On this scale, "0" indicates no pain, and "10" indicates the most severe pain imaginable.
Joint Range of Motion Evaluation | 3 times for 24 weeks
  During the assessments, three repeat measurements will be made using an electronic goniometer. For goniometric measurement, the pivot point will be placed on the lateral malleolus. The fixed arm will be kept parallel to the lateral midline of the fibula. The moving arm, on the other hand, will follow the lateral midline of the 5th metatarsal bone.
Tampa Kinesiophoby Scoring | 3 times for 24 weeks
  It is a 17-item scale developed to assess the fear of movement/re-injury. The lowest possible score on the test is 17; the highest score is 68; and a score higher than 37 is an indicator of poor health outcomes.
Star Excursion Test | 3 times for 24 weeks
  Physical performance that requires strength, flexibility, and proprioception is assessed through a dynamic test evaluating dynamic postural control and lower extremity injury risk associated with musculoskeletal injuries. The protocol of the test involves maintaining balance on the ipsilateral leg while reaching as far as possible with the contralateral leg.
Single Leg Stance Test | 3 times for 24 weeks
  Participants' standing balance will be assessed. Initially, one foot will be positioned on a firm and flat surface with the entire lower extremity in full extension, while the other lower extremity is positioned with the hip and knee flexed at 90 degrees. With their eyes closed, participants will start the timing when the foot not being tested loses contact with the ground, and the timing will stop when they place their foot back on the ground or when there is a significant increase in body sway.
The Side Hop Test | 3 times for 24 weeks
  It is a test that assesses the functional stability of patients. Patients will be asked to stand on one leg on the affected extremity. They will then be required to perform 10 jumps over two pre-determined strips that are spaced 30 cm apart.
Global Rating of Change Scale-GRC | 2 times for 52 weeks
  It will be used to evaluate patient satisfaction. It is designed to determine the amount of improvement or worsening of the patient over time.
  In our study, GRC consisting of 5 levels between -2 and +2 value ranges (-2: I am much worse, -1: I am worse, 0: I am the same, 1: I am better, 2: I am much better) was preferred.
Reproduction Test | 3 times for 24 weeks
  While the eyes of the individuals are closed, the ankle joints will be positioned and a goniometric measurement will be performed. Then, the patient will be brought to the starting position and asked to achieve the same movement. The difference between the two measurements will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Ayşenur Erekdağ, MSc, Principal Investigator — Bezmialem Vakif University
Locations (1):
- Acibadem Mehmet Ali Aydinlar University, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Background] Gribble PA, Bleakley CM, Caulfield BM, Docherty CL, Fourchet F, Fong DT, Hertel J, Hiller CE, Kaminski TW, McKeon PO, Refshauge KM, Verhagen EA, Vicenzino BT, Wikstrom EA, Delahunt E. Evidence review for the 2016 International Ankle Consortium consensus statement on the prevalence, impact and long-term consequences of lateral ankle sprains. Br J Sports Med. 2016 Dec;50(24):1496-1505. doi: 10.1136/bjsports-2016-096189. Epub 2016 Jun 3. PMID 27259753
- [Background] Owoeye OBA, Palacios-Derflingher LM, Emery CA. Prevention of Ankle Sprain Injuries in Youth Soccer and Basketball: Effectiveness of a Neuromuscular Training Program and Examining Risk Factors. Clin J Sport Med. 2018 Jul;28(4):325-331. doi: 10.1097/JSM.0000000000000462. PMID 29864071
- [Background] van Dijk CN, Vuurberg G. There is no such thing as a simple ankle sprain: clinical commentary on the 2016 International Ankle Consortium position statement. Br J Sports Med. 2017 Mar;51(6):485-486. doi: 10.1136/bjsports-2016-096733. Epub 2016 Oct 18. No abstract available. PMID 27797735
- [Background] Xue X, Ma T, Li Q, Song Y, Hua Y. Chronic ankle instability is associated with proprioception deficits: A systematic review and meta-analysis. J Sport Health Sci. 2021 Mar;10(2):182-191. doi: 10.1016/j.jshs.2020.09.014. Epub 2020 Oct 2. PMID 33017672
- [Background] Suttmiller AMB, McCann RS. Neural excitability of lower extremity musculature in individuals with and without chronic ankle instability: A systematic review and meta-analysis. J Electromyogr Kinesiol. 2020 Aug;53:102436. doi: 10.1016/j.jelekin.2020.102436. Epub 2020 Jun 1. PMID 32505988
- [Background] Needle AR, Lepley AS, Grooms DR. Central Nervous System Adaptation After Ligamentous Injury: a Summary of Theories, Evidence, and Clinical Interpretation. Sports Med. 2017 Jul;47(7):1271-1288. doi: 10.1007/s40279-016-0666-y. PMID 28005191
- [Background] Wilke J, Groneberg DA. Neurocognitive function and musculoskeletal injury risk in sports:A systematic review. J Sci Med Sport. 2022 Jan;25(1):41-45. doi: 10.1016/j.jsams.2021.07.002. Epub 2021 Jul 9. PMID 34303619